CLINICAL TRIAL: NCT01007227
Title: Achievement of Dietetic and Exercise Therapy Evaluated by Self-assessment Score Significantly Improved Endothelial Dysfunction in Patients With Metabolic Syndrome
Brief Title: Metabolic Syndrome and Fingertip Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Seigo Sugiyama, MD, PhD, Kumamoto University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 743EndothelialMetsyd
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle instruction (Other)
  Interventions: Other: Lifestyle instruction

INTERVENTIONS:
Other: Lifestyle instruction — Instruction dietetic and exercise therapy

SUMMARY:
Life-style intervention with dietetic and exercise therapy is an important fundamental approach to patients with metabolic syndrome (MetSyd) which may cause endothelial dysfunction leading to cardiovascular events. We investigated whether the life-style modification by dietetic and exercise instruction could improve endothelial dysfunction assessed by a new non-invasive and automatic device; digital reactive hyperemia peripheral arterial tonometry (RH-PAT).

DETAILED DESCRIPTION:
Outline of methods RH-PAT was measured in high-risk patients under 70 years old. The MetSyd was defined according to guidelines of the National Cholesterol Education Program Third Adult Treatment Panel (NCEP - ATP III). We instructed all MetSyd patients about the dietetic and exercise therapy according to the Japan Atherosclerosis Society Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases. we conducted a questionnaire survey of the self-assessment for dietetic and exercise instruction program, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Under 70 years old and preserved left ventricular systolic function (left ventricular ejection fraction ≥ 50%)

Exclusion Criteria:

* Severe valvular heart disease
* Atrial septal defect
* Myocarditis
* Cardiomyopathy
* Active inflammatory diseases
* Pulmonary hypertension
* Chronic kidney disease on hemodialysis
* Advanced hepatic disease
* Leukemia
* Schizophrenia; AND
* Cerebrovascular disease and residual hemiplegia.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Endothelial function assessed by RH-PAT | About 1 year later

SECONDARY OUTCOMES:
Metabolic status including waist circumference | About 1 year later

CONTACTS AND LOCATIONS:
Locations (1):
- Kumamoto University Hospital, Kumamoto, Kumamoto, Japan